CLINICAL TRIAL: NCT01013116
Title: A Double-blind Placebo-controlled Trial to Evaluate Efficacy and Safety of Specific Subcutaneous Immunotherapy in Patients With Perennial Allergic Rhinitis Due to House Dust Mites
Brief Title: Evaluation of Efficacy and Safety of Specific Immunotherapy With Modified Allergen Extracts of House Dust Mites
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Roxall Medizin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SBC-2009-002B
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- modified allergen extract of house dust mites (Experimental)
  Interventions: Biological: modified allergen extract of house dust mites
- Placebo (Placebo Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: modified allergen extract of house dust mites — subcutaneous injections
  Arms: modified allergen extract of house dust mites
Biological: placebo — subcutaneous injections
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of specific subcutaneous immunotherapy with modified allergen extracts.

ELIGIBILITY:
Inclusion Criteria:

* Positive history of perennial allergic rhinitis due to house dust mites
* Positive screening skin prick test (wheal diameter > 3 mm)
* Compliance and ability of the patient to complete a Diary Card for self-evaluating of the symptoms and antisymptomatic medication
* Signed and dated patient´s Informed Consent,

Exclusion Criteria:

* Previous immunotherapy with mite extracts within the last 3 years,
* Simultaneous participation in other clinical trials,
* Other reasons contra-indicating an inclusion into the trial according to the investigator´s estimation (e.g. poor compliance),
* Auto-immune disorders,
* Severe chronic inflammatory diseases,
* Malignancy,
* Alcohol abuse,
* Existing or intended pregnancy, lactation and/or lack of adequate contraceptive protection,
* Treatment with beta-blockers (incl. local application) and/or other contra-indicated drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Symptom and medication score | 1 year

SECONDARY OUTCOMES:
Safety of the treatment | 1 year
Documentation of adverse events | 1 year
Clinical global improvement | 1 year
Quality of Life Questionnaire | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Madrid, Spain